CLINICAL TRIAL: NCT06933589
Title: Effect of a New Optimized Plant Ingredient on the Plant Protein of Seniors at Cardio-metabolic Risk - P-Probs Project
Brief Title: Effect of a New Optimized Plant Ingredient on the Plant Protein of Seniors at Cardio-metabolic Risk
Acronym: P-Probs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: RBHP 2023 RICHARD; 2023-A00959-36 (Other: ANSM)
Record Dates: First submitted 2024-09-03; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-09

CONDITIONS: Nutrition, Healthy; Metabolic Syndrome
Keywords: Protein
MeSH Terms: conditions — Metabolic Syndrome | interventions — Plant Proteins; Milk Proteins

STUDY DESIGN:
Intervention Model Description: Each subject is asked to test 2 different products during 2 kinetics of 9.5 hours each. Each kinetic is separated by a wash-out period of at least 2 weeks.
Who Masked: Care Provider
Masking Description: Participants will not know which protein ingredient is included in the test-meal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plant proteins (Experimental): Test meal incorporating an optimized plant protein ingredient
  Interventions: Other: Test meal with plant protein
- Milk protein (Active Comparator): Test meal incorporating milk proteins
  Interventions: Other: Test meal with milk protein

INTERVENTIONS:
Other: Test meal with plant protein — The plant protein blend is made up of 5 protein ingredients for which the food grade is guaranteed: a rice protein isolate, a potato protein isolate, a lupin protein isolate, a corn protein isolate.
  Arms: Plant proteins
Other: Test meal with milk protein — The milk protein product is a food-grade protein isolate.
  Arms: Milk protein

SUMMARY:
The aim of the study is to compare the use of amino acids in whole-body protein metabolism in elderly consumers at risk of metabolic syndrome, after ingestion of 2 foods differing only in the nature of their proteins (optimized blend of vegetable proteins versus milk proteins).

The protocol consists in studying the postprandial evolution of protein metabolism. Two products will be tested: one based on dairy proteins, the other on an optimized blend of vegetable proteins).

DETAILED DESCRIPTION:
Written consent will be obtained from subjects after they have been informed of the aims, nature and possible risks of the study.

Prior to inclusion, subjects will have a medical check-up carried out in the Nutritional Exploration Unit (UEN), including an interview about personal and family history and medication taken, as well as a standard medical examination and a blood test for a biological work-up (9.5 ml). Compliance with inclusion/exclusion criteria will be verified during this examination.

Subjects included in the study will come to the UEN to undergo the pre-study dietary visit and to complete the two study days of 9.5 hours each, at least two weeks apart.

For each study day, volunteers will arrive in the morning with an empty stomach. Two vascular catheters will be implanted. One catheter will provide continuous intravenous infusion of a labelled amino acid (13C Leucine) for a total duration of 9.5 hours. The second catheter will be used for blood sampling (8 ml), performed on an empty stomach and then, kinetically after ingestion of one of the two study products, in the form of food prepared on site. The IV-infused tracers will be used to monitor the kinetics of leucine appearance in plasma, and to quantify amino acid utilization flows at whole-body level (protein synthesis, degradation). Blood samples will also be taken to determine aminoacidemia, glycemia, insulinemia and plasma concentrations of hormones involved in regulating food intake (grelin, cholecystokinin, Glucagon-like-peptide-1 (GLP1), peptide YY (PYY).

Exhaled gases will be collected during the study days. Indirect calorimetry measurements lasting 20 minutes will be taken in the post-absorptive and post-prandial periods. Seven indirect calorimetry measurements will be taken on each study day. Finally, subjects will be asked to rate their satiety on a visual analog scale, at different times during the study days.

Subjects will also be asked to complete a tolerance questionnaire on each study day.

At the end of each study day, volunteers will have a snack at the study center before their departure. Any intercurrent events will be recorded in the observation notebook.

Allocation of the product sequence to subjects will be carried out by a random draw (generation of a random list) before the start of the study.

The volume of blood drawn per volunteer is 128 ml/study day, to which must be added 9.5 ml for the biological screening test, i.e. 265.5 ml for the entire study.

During the 3 days preceding each study day, the subjects' protein intake will be monitored. Standard menus were proposed, providing 1.2 g protein/kg/d. The meal on the evening before each study day will be standardized and identical for each day. To check compliance with the dietary instructions, volunteers will complete a dietary record for the 3 days preceding each study day.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference > 94cm
* Triglycerides > 1.5 g/L or HDL cholesterol < 0.4 g/L
* Fasting blood glucose < 1.26g/L
* Biological profile considered compatible with study participation,
* Venous status judged satisfactory by the nurses, allowing catheter placement for the study,
* Individuals able to sign the informed consent form,
* Persons subject to a social security scheme.

Exclusion Criteria:

* Subjects on special diets (vegetarian, vegan, etc.),
* Subject showing a weight loss ≥ 5% in 1 month or ≥ 10% in 6 months compared to usual weight.
* Subject refusing to stop taking dietary supplements for the duration of the study,
* Subject refusing to consume any of the proposed products,
* Subject with food allergy(ies) to one or more components of the products under study, or with a contraindication to the consumption of these products,
* Subjects with a pathology or treatment (antidiabetics, hypolipidemics, corticoids, neuroleptics) judged by the investigator to be incompatible with the study,
* Subjects with dysthyroidism that has not been stabilized for at least 3 months,
* Subject with unstabilized hypertension for at least 3 months,
* Subject with a medical and/or surgical history deemed by the investigator to be incompatible with the trial,
* Subject having undergone surgery that could interfere with the study objectives (as judged by the investigating physician) in the 3 months preceding the study,
* Smoking > 5 cigarettes/day,
* Alcohol > 3 glasses/day,
* Claustrophobic subject,
* Person refusing to be registered with the French Ministry of Health's Fichier National des Volontaires Sains,
* Major under guardianship or with limited rights,
* Subject not affiliated to social security,
* Subject in a period of exclusion from a previous study or having received a total amount of compensation exceeding 6000 euros over the 12 months preceding the start of the trial (after verification in the Fichier des Volontaires pour la Recherche Biomédicale).

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-14 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Whole body protein metabolism | 8 months (including mass spectrometry analysis and calculations)
  Body leucine flux kinetics: oxidation, protein synthesis

SECONDARY OUTCOMES:
Satiety effect | 12 months
  Satiety-enhancing effect of proteins, assessed using a visual analog scale
Evolution of blood parameters related to satiety | 12 months
  Plasma concentrations of glucose, insulin, ghrelin, cholecystokinin, glucagon-like-peptide (GLP1), peptide YY (PYY) and amino acids
Product tolerance | 12 months
  Product tolerance assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Principal Investigator — University Hospital, Clermont-Ferrand; Didier REMOND, Study Director — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France